CLINICAL TRIAL: NCT03648346
Title: A Dose Block-randomized, Double Blind, Placebo Controlled, Dose-escalation Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics After Multiple Dosing of HL217 Eye Drop in Healthy Male Subjects
Brief Title: A Dose-escalation Clinical Trial After Multiple Dosing of HL217 Eye Drop in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: HL217-102
Record Dates: First submitted 2018-06-19; First posted 2018-08-27 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: HL217 Ophathalmic Solution BID (Experimental): Low dose: two drops of 3 mg/mL of the treatment in one eye twice a day
  Interventions: Drug: Cohort 1: HL217 Ophathalmic Solution BID
- Cohort 2: HL217 Ophathalmic Solution QID (Experimental): High dose: two drops of 3 mg/mL of the treatment in one eye 4 times a day
  Interventions: Drug: Cohort 2: HL217 Ophathalmic Solution QID
- Placebo Ophathalmic Solution (Placebo Comparator): Placebo: two drops of placebo in one eye twice a day or 4 times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cohort 1: HL217 Ophathalmic Solution BID — Two drops of 3 mg/mL of the treatment in one eye twice a day
  Other Names: 3mg/mL
  Arms: Cohort 1: HL217 Ophathalmic Solution BID
Drug: Cohort 2: HL217 Ophathalmic Solution QID — Two drops of 3 mg/mL of the treatment in one eye 4 times a day
  Other Names: 3mg/mL
  Arms: Cohort 2: HL217 Ophathalmic Solution QID
Drug: Placebo — Placebo eye drops
  Arms: Placebo Ophathalmic Solution

SUMMARY:
The study is a single center, double-blind, randomized, parallel group, multiple ascending dose study in 16 healthy male volunteers. Subjects will receive multiple eye drop doses during 14 days of the treatment (HL217 or placebo according to the randomization). There will be 2 cohorts of 8 subjects (6 HL217 vs 2 placebo) receiving the following doses:

* Cohort 1 : two drops of 3 mg/mL of the treatment in one eye twice a day (low dose),
* Cohort 2 : two drops of 3 mg/mL of the treatment in one eye 4 times a day (high dose).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of HL217 after multiple eye drop administrations at different doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, aged between 18 and 50 years inclusive
2. Non-smoker subject or smoker of not more than 10 cigarettes a day and able to stop smoking 24 hour prior to admission until discharge
3. Body weight ≥ 50 kg and BMI between 18 and 30 kg/m²
4. Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination) including complete ocular examination
5. Normal Blood Pressure (BP) and Heart Rate (HR) after 10 minutes in supine position:

   * 90 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 140 mmHg,
   * 45 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
   * 40 bpm ≤ HR ≤ 100 bpm,
   * Or considered NCs by investigators;
6. Normal ECG recording on a 12-lead ECG:

   * 120 < PR < 200 ms,
   * QRS < 120 ms,
   * QTcf ≤ 430 ms,
   * No sign of any trouble of sinusal automatism,
   * Or considered NCs by investigators;
7. Laboratory parameters within the normal range of the laboratory (haematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator
8. Normal dietary habits
9. Signing a written informed consent prior to selection
10. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurologic, psychiatric, systemic, infectious or ocular disease
2. Frequent headaches and / or migraine, recurrent nausea and / or vomiting
3. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20 mmHg within two minutes when changing from the supine to the standing position
4. Blood donation (including in the frame of a clinical trial) within 2 months before administration or apheresis within 20 days before administration
5. General anaesthesia within 3 months before administration
6. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician (including allergy to fluorescein)
7. Inability to abstain from intensive muscular effort;
8. No possibility of contact in case of emergency;
9. Any drug or herbal medicine intake (except paracetamol) during the last 14 days prior to the first administration, any over the counter medicine or vitamin during the last 7 days prior to the first administration
10. Subjects who have taken drug metabolizing enzyme inducing agents and inhibitors such as barbitals within a month prior to the first administration
11. History or presence of drug or alcohol abuse (alcohol consumption > 30 grams / day);
12. Excessive consumption of beverages with xanthine bases (> 5 cups or glasses / day) and not able to stop 24h prior to admission until discharge
13. Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2
14. Major surgery (general or ocular) within 28 days prior to randomization or major surgery planned during the next 6 months
15. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development
16. Subjects within an exclusion period of a previous study or subjects who have taken any investigational product from other clinical trials within 60 days from the start of the study (from the administration of investigational product)
17. Subjects with an allergy to Fluorescein
18. Subjects with previous participation in the current study
19. Subject under administrative or legal supervision
20. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Clinical parameter: Adverse Events (AE) | Day 1 (Pre-dose) to Day 22 (End of study visit)
  AEs will be coded according to the MedDRA. They will be classified into pre-defined standard categories according to chronological criteria
Clinical parameter: Physical examination | Day -1, Day 1 (Before administration, 4h, 8h, 12h), Day 2 (24h), Day 3 to 15, Day 22 (End of study visit)
  Physical examination recorded during the study will be individually listed and quantitative parameters will be summarized by using descriptive statistics
Clinical parameter: Vital signs | Day -1, Day 1 (Before administration, 4h, 8h, 12h), Day 2 (24h), Day 3 to 15, Day 22 (End of study visit)
  Vital signs recorded during the study will be individually listed and quantitative parameters will be summarized by using descriptive statistics
Clinical parameter: ECG (ElectroCardioGram) | Day -1, Day 1 (Before administration), Day 2, Day 15, Day 22 (End of study visit)
  ECG recorded during the study will be individually listed and quantitative parameters will be summarized by using descriptive statistics
Clinical parameter: Laboratory parameters | Day -1, Day 2, Day 15, Day 22 (End of study visit)
  All laboratory values recorded during the study will be individually listed and flagged for values outside reference ranges and for clinical relevance (assessed by investigator)
Local tolerance test | Day -1, Day 1 (Before administration, 4h, 8h, 12h), Day 2 (24h), Day 3 to 15, Day 22 (End of study visit)
  Redness, tingling and others should be checked

SECONDARY OUTCOMES:
Pharmacokinetic assessments: Cmax | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  observed maximum plasma concentration of HL217
Pharmacokinetic assessments: Tmax | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  first time to reach Cmax
Pharmacokinetic assessments: AUCt | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  area under the plasma concentration curve from administration up to the last quantifiable concentration at time t
Pharmacokinetic assessments: AUCinf | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  area under the plasma concentration-time curve from administration up to infinity with extrapolation of the terminal phase
Pharmacokinetic assessments: Kel | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  elimination rate constant
Pharmacokinetic assessments: t1/2 | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  plasma elimination half-life
Pharmacokinetic assessments: %AUCextra | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  percentage of extrapolated AUCinf
Pharmacokinetic assessments: Vd/F | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  volume of distribution
Pharmacokinetic assessments: CL/F | 0h, 12h, 12h05min, 12h15min, 12h30min, 12h45min, 13h, 14h, 15h, 16h, 18h, 20h, 24h, 28h and 32hours after the last administration at Day 14
  Clearance

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, M.D, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins OPTIMED, Gières, France